CLINICAL TRIAL: NCT05255146
Title: Cryoanalgesia and Post-thoracotomy Pain in Minimally Invasive Cardiothoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00113974
Record Dates: First submitted 2022-01-31; First posted 2022-02-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cryotherapy Effect; Post Operative Pain
Keywords: Minimally Invasive cardiac surgery; cryoanalgesia; mitral valve surgery; ASD repair; thoracotomy; pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized, double-blinded, placebo-controlled trial evaluating the effect of intercostal cyroablation on the development of post-thoracotomy pain. With the use of computer-generated randomized blocks, patients will be assigned to either Cryoanalgesia or no-cryoanalgesia before undergoing surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized to either study group before surgery without the patient's knowledge of which group they are in. The surgeons (care providers) will need to be aware of the intervention so that they can supply the cryoanalgesia or not peri-operatively. The investigator and data analyst will also be blind to the intervention type when collecting patient outcome information and doing statistical analysis. Randomization will be documented in secure password protected databases that only the surgeons will have access too, matching patient identifiers to intervention groups for reference for final data presentation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Cryoanalgesia (Experimental): Patients receiving cryoanalgesia peri-operatively during minimally invasive cardiothoracic surgery
  Interventions: Device: Atricure Inc. Nitrous oxide Cryoprobe
- Control Group: No Cyroanalgesia (No Intervention): Patients receiving minimally invasive cardiothoracic surgery who do not receive cryoanalgesia.

INTERVENTIONS:
Device: Atricure Inc. Nitrous oxide Cryoprobe — Cryoanalgesia will be given by applying a nitrous oxide-cooled probe (AtriCure, Inc. 2000) locally to intercostal nerves in the 4th, 5th, and 6th rib spaces after completion of the surgical repair and before surgical closure. The probe will be cooled to -60°C and held on each location for 60 sec.
  Arms: Intervention Group: Cryoanalgesia

SUMMARY:
Minimally invasive cardiothoracic surgery is often associated with chronic pain syndrome, out of keeping with the extent of surgical dissection. This is thought to be because of damage to the intercostal nerves by compression and traction by the surgical equipment. Cryoanalgesia is long-standing technique that freezes nerves locally to temporarily block pain sensation, which is currently used to treat acute post-operative pain in lung dissections and the Nuss procedure. We intend to perform a trial to assess whether using cryoanalgesia on intercostal nerves intraoperatively, reduces post-operative pain following minimally invasive cardiothoracic surgery.

DETAILED DESCRIPTION:
Objective:

To characterize the effects of peri-operative intercostal cryoablation for the prevention of post thoracotomy pain following minimally invasive mitral valve surgery or atrial septal defect repair.

Rationale:

Minimally invasive cardiothoracic surgery is often associated with prolonged post-operative neuropathic pain not consistent with the acute pain experience of the initial surgery [1]. This is often thought to be secondary to an intercostal neuralgia caused by traction injuries to the intercostal neurovascular bundles by the surgical ports, a mini-thoracotomy, and mechanical retraction of the ribs.

Cryoanalgesia is an older but clinically relevant technique that causes local destruction of nerve axons using a nitrous oxide-cooled probe to -60°C [2]. This allows for temporary acute pain relief without damaging the endoneurium, allowing the peripheral nerves to regrow post-operatively. Previous studies have demonstrated cryoanalgesia as having improved acute post-operative pain vs opioids alone or similar acute pain management vs epidural analgesia [3,4]. A few studies have assessed Cryoanalgesia in thoracic surgery patients; however, these studies have focused primarily on lung operations involving pulmonary resections, and did not include cardiac operations [5,6]. Furthermore, studies that evaluated cardiothoracic operations specifically, were either retrospective or prospective in approach and did not include a representative variety of cardiac operations [7-9]. Therefore, we hope that by using intercostal cryoablation in minimally invasive cardiac surgery patients, we might improve post-operative pain and reduce analgesic requirements.

Sample Size and Statistical Considerations:

Analyses will be conducted on an intention-to-treat basis. Relative and absolute risk will be calculated with respect to the primary and secondary outcomes. We calculate a sample size of 50 patients per group in order to detect a reduction in incidence of post-thoracotomy pain from 50% to 20% (α=0.05, power=0.8). This includes an anticipated rate of non-completion of 15%.

Expected Results:

Based on our hypotheses and previous human RCT's, we expect intercostal cryoablation to improve post-thoracotomy pain when compared to controls. Furthermore, we expect an improvement in our secondary outcomes including sleep quality and analgesic requirements. Cryoanalgesia's efficacy in acute post-operative pain management is well documented in the neuropathic pain literature and has been used in a number of clinical trials. We hope that applying this concept to minimally invasive cardiothoracic procedures, we can see similar results in improved post-thoracotomy pain as reported by previous studies. We believe that, if successful, this project will offer an alternative and improved pain management regimen for patients undergoing minimally invasive thoracic surgery.

Significance:

The study proposed aims to provide new insight into the management of neuropathic pain associated with minimally invasive thoracic surgery. Pain -whether acute, chronic, nociceptive, or neuropathic- creates a significant burden to the patient, as well as to those around them. Our ultimate aim is to limit the overall pain experienced by patients. In doing this, we hope to influence a multitude of factors that affect patient welfare, including mood, patient safety, return to independence, return to work, etc. Many of these factors are often much more subjective and difficult to capture within the analytical framework of a clinical trial. However, it is our hope that by reducing pain, itself, we can continue to improve patient satisfaction and consequently, patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older scheduled for elective minimally invasive mitral valve surgery or atrial septal defect repair.

Exclusion Criteria:

* Patients will be excluded if they are unable to fill in detailed health and pain related questionnaires, psychiatric disease preventing recall or accurate descriptions of pain, chronic pain syndromes, alcohol or illegal substance abuse, or pregnancy. Exclusion criteria also includes chronic use of opioids, allergy to morphine, bupivacaine, and/or ibuprofen, average pain during the last week >4 on a numerical rating scale from 0 to 10 with 0 indicating "no pain" and 10 indicating "the worst pain imaginable", contraindications to thoracic epidurals, prior chest surgery, or participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain Day 1 | 1 day post-op
  The incidence of significant post-thoracotomy pain will be assessed by the Brief Pain Inventory, asked in-person by one of the researchers.
Post-operative Pain Day 3 | 3 days post-op
  The incidence of significant post-thoracotomy pain will be assessed by the Brief Pain Inventory, asked in-person by one of the researchers.
Post-operative Pain Day 5 | 5 days post-op
  The incidence of significant post-thoracotomy pain will be assessed by the Brief Pain Inventory, asked in-person by one of the researchers.
Long-term Post-operative Pain | 6 weeks post-op
  The incidence of significant post-thoracotomy pain will be assessed by the Brief Pain Inventory by asking the participants via phone call.

SECONDARY OUTCOMES:
Sleep Quality | 1 week post-op
  Average sleep quality will be assessed by asking participants to rate their sleep over the first post-operative that they spent in-hospital. This will be scored numerically from 0 to 10, with 0 indicating extremely poor sleep quality and 10 indicating extremely good sleep quality.
Consumptions of Analgesics Day 1 | 1 day post-op
  Average daily consumption of analgesics, adjusted to morphine equivalents, will be collected from patient chart information while they are admitted.
Consumptions of Analgesics Day 3 | 3 days post-op
  Average daily consumption of analgesics, adjusted to morphine equivalents, will be collected from patient chart information while they are admitted.
Consumptions of Analgesics Day 5 | 5 Days post-op
  Average daily consumption of analgesics, adjusted to morphine equivalents, will be collected from patient chart information while they are admitted.
Long-term Consumptions of Analgesics | 6 weeks post-op
  Average daily consumption of analgesics, adjusted to morphine equivalents, over the 7 days prior to assessment.
Length of Hospital Stay | approximately 2 weeks post-op
  Hospital length of stay, measured in days, will be determined by their discharge date post-operatively and their date of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Abeline R Watkins, BSc, Principal Investigator — UofA Research/Department of Cardiac Surgery; Andrew O'Connell, MD, Principal Investigator — UofA Department of Cardiac Surgery

REFERENCES:
- [Background] Guastella V, Mick G, Soriano C, Vallet L, Escande G, Dubray C, Eschalier A. A prospective study of neuropathic pain induced by thoracotomy: incidence, clinical description, and diagnosis. Pain. 2011 Jan;152(1):74-81. doi: 10.1016/j.pain.2010.09.004. Epub 2010 Nov 13. PMID 21075523
- [Background] Muller LC, Salzer GM, Ransmayr G, Neiss A. Intraoperative cryoanalgesia for postthoracotomy pain relief. Ann Thorac Surg. 1989 Jul;48(1):15-8. doi: 10.1016/0003-4975(89)90169-0. PMID 2764595
- [Background] Ju H, Feng Y, Yang BX, Wang J. Comparison of epidural analgesia and intercostal nerve cryoanalgesia for post-thoracotomy pain control. Eur J Pain. 2008 Apr;12(3):378-84. doi: 10.1016/j.ejpain.2007.07.011. Epub 2007 Sep 17. PMID 17870625
- [Background] Park R, Coomber M, Gilron I, Shanthanna H. Cryoanalgesia for postsurgical pain relief in adults: A systematic review and meta-analysis. Ann Med Surg (Lond). 2021 Aug 5;69:102689. doi: 10.1016/j.amsu.2021.102689. eCollection 2021 Sep. PMID 34408872
- [Background] Brichon PY, Pison C, Chaffanjon P, Fayot P, Buchberger M, Neron L, Bocca A, Verdier J, Sarrazin R. Comparison of epidural analgesia and cryoanalgesia in thoracic surgery. Eur J Cardiothorac Surg. 1994;8(9):482-6. doi: 10.1016/1010-7940(94)90019-1. PMID 7811482
- [Background] Sepsas E, Misthos P, Anagnostopulu M, Toparlaki O, Voyagis G, Kakaris S. The role of intercostal cryoanalgesia in post-thoracotomy analgesia. Interact Cardiovasc Thorac Surg. 2013 Jun;16(6):814-8. doi: 10.1093/icvts/ivs516. Epub 2013 Feb 19. PMID 23424242
- [Background] Tanaka A, Al-Rstum Z, Leonard SD, Gardiner BD, Yazij I, Sandhu HK, Miller CC 3rd, Safi HJ, Estrera AL. Intraoperative Intercostal Nerve Cryoanalgesia Improves Pain Control After Descending and Thoracoabdominal Aortic Aneurysm Repairs. Ann Thorac Surg. 2020 Jan;109(1):249-254. doi: 10.1016/j.athoracsur.2019.07.083. Epub 2019 Sep 12. PMID 31521592
- [Background] Clemence J Jr, Malik A, Farhat L, Wu X, Kim KM, Patel H, Yang B. Cryoablation of Intercostal Nerves Decreased Narcotic Usage After Thoracic or Thoracoabdominal Aortic Aneurysm Repair. Semin Thorac Cardiovasc Surg. 2020 Autumn;32(3):404-412. doi: 10.1053/j.semtcvs.2020.01.008. Epub 2020 Jan 20. PMID 31972300
- [Background] Bucerius J, Metz S, Walther T, Doll N, Falk V, Diegeler A, Autschbach R, Mohr FW. Pain is significantly reduced by cryoablation therapy in patients with lateral minithoracotomy. Ann Thorac Surg. 2000 Sep;70(3):1100-4. doi: 10.1016/s0003-4975(00)01766-5. PMID 11016387
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870